CLINICAL TRIAL: NCT03057743
Title: Imaging of in Vivo Sigma-2 Receptor Expression With 18F-ISO-1 Positron Emission Tomography in Metastatic Breast Cancer
Status: Terminated | Type: Observational
Why Stopped: Difficulty enrolling subjects
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 03116
Record Dates: First submitted 2017-02-16; First posted 2017-02-20 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: METASTATIC BREAST CANCER
MeSH Terms: conditions — Breast Neoplasms | interventions — Positron-Emission Tomography; Positron Emission Tomography Computed Tomography; Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Positron emission tomography (PET/CT) imaging
Device: radiotracer [18F]ISO-1

SUMMARY:
Pilot study using [18F]ISO-1 PET/CT to image sigma-2 receptor binding in metastatic breast cancer. Correlate baseline uptake and change in uptake after therapy with time to progression and standard and experimental pathology assays of biopsy or surgical tissue. The target population is up to 30 adult patients at least 18 years, with at least one site of disease outside the liver by at least one type of standard imaging.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Biopsy proven or clinically documented metastatic breast cancer with at least one lesion outside the liver by standard imaging (e.g. CT, MRI, Bone Scan, Ultrasound, FDG PET/CT)
* Plan to start new systemic therapy for metastatic disease.
* Participants must be informed of the investigational nature of this study and be willing to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria:

* Females who are pregnant at the time of screening will not be eligible for this study, urine or serum pregnancy test will be performed in women of child-bearing potential at the time of screening.
* Inability to tolerate imaging procedure in the opinion of an investigator or treating physician.
* Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metastatic Breast Cancer
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2016-04-05 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth MdDonald, MD, Ph.D, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States